CLINICAL TRIAL: NCT04488666
Title: A Clinical Evaluation of a Novel, Single-Use, Negative Pressure Wound Therapy (NPWT) System for the Management of Closed Surgical Wounds
Brief Title: Clinical Evaluation of a Novel Incisional NPWT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aatru Medical LLC (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Surgical Wound
Keywords: incisional NPWT
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- npSIMS (Experimental): Group will receive the Aatru Medical npSIMS device
  Interventions: Device: npSIMS

INTERVENTIONS:
Device: npSIMS — incisional NPWT
  Other Names: negative pressure Surgical Incision Management system

SUMMARY:
A study of the first clinical use in humans of a novel NPWT system (npSIMS) to assess the suitability, safety and efficacy of the system for the management of closed surgical wounds

DETAILED DESCRIPTION:
The purpose of this investigation is to test the functionality of a novel, non-electric NPWT device: npSIMS (negative pressure Surgical Incision Management System) from Aatru Medical LLC (Ohio, USA) which uses an exothermic chemical process to extract the oxygen from the air contained within the dressing (air contains 21% O2) and hence bring and maintain the system to between -160 and -80 mmHg below atmospheric pressure (760 mmHg). The dressing and the chemical reaction pump module can be manufactured for significantly less than the cost of electromechanical NPWT systems and can be profitably marketed at a discount to the cost of existing commercial devices. The Aatru Medical NPWT system could transform the economics and increase the availability of this therapy across the world.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female ≥ 18 years of age 2. Participant will undergo an elective sternotomy, thoracotomy, caesarean section (C-section) or skin surgery incision with closure by sutures or staples 3. Participant will undergo a surgical procedure resulting in a closed approximately linear incision between 5 cm and 13 cm in length inclusive so that the npSIMS dressing covers the wound with a minimum of 1 cm overlap at each end 4. Participant is willing and able to take part in the study and provide written informed consent.

-

Exclusion Criteria:

1. Participants will undergo post-surgical radiotherapy or chemotherapy
2. Participants who, in the opinion of the Investigator, have an existing health condition that would compromise their participation and follow-up in this study
3. Participant will undergo emergency surgery
4. Participant is sensitive to or known to have allergies to silicone/acrylic adhesives
5. Participant has malignancy in the wound bed or margins of the wound
6. Participant has wound with confirmed and untreated osteomyelitis
7. Participant has wound with non-enteric and unexplored fistulas
8. Participant has wound with necrotic tissue with eschar present
9. Participant has exposed arteries, veins, nerves or organs
10. Participant has exposed anastomotic sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Mean (median) number of days of negative pressure delivered to the incision up to day 7 | 7 days
  To assess the maintenance and reliability with which negative pressure is delivered for the 7-day NPWT period.

SECONDARY OUTCOMES:
Mean (median) clinician assessment of exudate management on 5-point Numerical Rating Score (NRS) at day 7 ±2 and at any npSIMS replacement. | 7 Days
  5 is excellent exudate management; 4 is good; 3 is adequate; 2 is poor; 1 is inadequate
Mean (median) days wear time of the adhesive dressing up to day 7 | 7 days
  To assess the wear time of the adhesive dressing
Mean (median) days longevity of the chemical vacuum source up to day 7 | 7 Days
  To assess the longevity of the chemical vacuum source
Presence or absence of blisters on day 7 ±2 | 7 days
  Condition of the peri wound skin
Mean (median) overall observer and participant scores in the POSAS - Patient Observer Scar Assessment Scale on day 14 ±2 clinic follow up. | 14 days
  To assess the appearance of the closed incision and scar. Each item of the POSAS is rated on a 10-point score. The lowest score is '1', which corresponds to the situation of normal skin (i.e. normal pigmentation, no itching). Score 10 equals the largest difference from normal skin (i.e. the worst imaginable scar or sensation)
Frequency of surgical wound complications according to the ASEPSIS wound score at day 14 ±2 clinic and day 30±2 remote follow up. | 30 Days
  Assess the Frequency of Surgical site infections. A higher ASEPSIS score indicates impaired wound healing (a score of >10 indicates an increasing probability and severity of infection)
Mean (median) wound pain score using a 0 -10 NRS (numerical rating score) by the study participant each day up to day 7±2. 10 is worst imaginable pain; 0 is no pain. | 7 days
  To assess wound pain daily in the 7 day post-operative period
Frequency of adverse events (non-device related, and device related) up to day30 ±2 | 30 Days
  To assess the occurrence of adverse events
Mean (median) ease of use score from patients on 5-point NRS (numerical rating score) assessed at day 7 ±2. 5 is excellent ease of use; 4 is good; 3 is adequate; 2 is poor; 1 is inadequate | 7 days To assess the ease of use by patients assessments
  To assess the ease of use by patients assessments
Mean (median) ease of use score from clinicians on 5-point NRS (numerical rating score) assessed at day 7 ±2. 5 is excellent ease of use; 4 is good; 3 is adequate; 2 is poor; 1 is inadequate | 7 days
  To assess the ease of use by clinicians assessments
Mean (median) score of overall clinician acceptability of the NPWT system (pump & dressing) on 5-point NRS assessed at day 14 ±2. 5 is Excellent incision management system; 4 is good; 3 is adequate; 2 is poor; 1 is inadequate | 14 days
  To assess overall clinician acceptability of the NPWT system

CONTACTS AND LOCATIONS:
Overall Officials: Jon Mathy, MD, Principal Investigator — 1Auckland Regional Plastic Surgery Unit and University of Auckland School of Medicine
Locations (1):
- Middlemore Clinical Trials, Auckland, New Zealand